CLINICAL TRIAL: NCT00986115
Title: Efficacy and Safety of the Use of Memantine for Preserving Cognition in Adult Patients With Epilepsy
Acronym: Forest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: our site was unable to enroll any qualified subjects
Sponsor: University of California, Davis (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 200816572
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
Keywords: epilepsy; memory; cognition; memantine
MeSH Terms: conditions — Epilepsy | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Active Comparator): After a two-month prospective baseline during which seizure frequency and neurocognitive parameters are documented, patients will be randomized to either memantine or placebo and evaluated after twelve months on study drug. The treatment period will consist of a one month dose escalation phase, followed by an eleven month maintenance phase. The dose escalation is 5 mg in PM for days 1-7, 5 mg twice daily for days 8-14, 5 mg in AM and 10 mg in PM for days 15-21 and 10 mg twice daily from day 22 and continue.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): After a two-month prospective baseline during which seizure frequency and neurocognitive parameters are documented, patients will be randomized to either memantine or placebo and evaluated after twelve months on study drug. The treatment period will consist of a one month dose escalation phase, followed by an eleven month maintenance phase. The dose escalation is 5 mg in PM for days 1-7, 5 mg twice daily for days 8-14, 5 mg in AM and 10 mg in PM for days 15-21 and 10 mg twice daily from day 22 and continue.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — After a two-month prospective baseline during which seizure frequency and neurocognitive parameters are documented, patients will be randomized to either memantine or placebo and evaluated after twelve months on study drug. The treatment period will consist of a one month dose escalation phase, followed by an eleven month maintenance phase. The dose escalation is 5 mg in PM for days 1-7, 5 mg twice daily for days 8-14, 5 mg in AM and 10 mg in PM for days 15-21 and 10 mg twice daily from day 22 and continue.
  Other Names: Namenda; Axura
  Arms: Memantine
Drug: Placebo — After a two-month prospective baseline during which seizure frequency and neurocognitive parameters are documented, patients will be randomized to either memantine or placebo and evaluated after twelve months on study drug. The treatment period will consist of a one month dose escalation phase, followed by an eleven month maintenance phase. The dose escalation is 5 mg in PM for days 1-7, 5 mg twice daily for days 8-14, 5 mg in AM and 10 mg in PM for days 15-21 and 10 mg twice daily from day 22 and continue.
  Arms: Placebo

SUMMARY:
People with epilepsy often experience problems with their memories and other thinking skills that get worse over time. The investigators hope to learn more about whether a drug called memantine can help improve or stabilize (keep the same) memory and other thought processes in people with epilepsy by blocking a chemical that is released in the brain during seizures. The investigators also want to see if memantine changes the frequency (how often) people with epilepsy have seizures. Memantine is currently approved by the United States Food and Drug Administration (FDA) for treatment of patients with Alzheimer's disease.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled trial of the effects of memantine in adult epilepsy patients. Patients will be assessed for neurocognitive outcomes, seizure frequency and side effects. After a two-month prospective baseline during which seizure frequency and neurocognitive parameters are documented, patients will be randomized to either memantine or placebo and evaluated after twelve months on study drug. The treatment period will consist of a one month dose escalation phase, followed by an eleven month maintenance phase. The dose escalation is 5 mg in PM for days 1-7, 5 mg twice daily for days 8-14, 5 mg in AM and 10 mg in PM for days 15-21 and 10 mg twice daily from day 22 and continue. The neuropsychological battery performed during baseline will be repeated at the end of the twelve month treatment period. No special procedures are required for this study, except the neuropsychological testing, which is not a routinely performed evaluation for adult epilepsy outpatients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with temporal lobe epilepsy, aged 18-65
2. Seizure frequency of less than three per month
3. Stabilized treatment for epilepsy, including AEDs and vagus nerve stimulation
4. Intelligence Quotient of >70
5. Native English speaker (most of the neuropsychological/cognitive tests have yet to be translated and/or validated in non-English speaking populations. Thus, at this point we are limited to testing English speakers, only.)
6. Able to count seizures accurately and maintain a seizure diary
7. Recent AED levels performed within the last month within therapeutic range

Exclusion Criteria:

1. Progressive neurologic disease
2. Severe medical illness, including renal insufficiency
3. Severe depression, bipolar disease or psychosis
4. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference in neuropsychological test scores over time between memantine and placebo treated groups of temporal lobe epilepsy patients. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rogawski, MD, PhD, Principal Investigator — University of California, Davis Health System
Locations (1):
- University of California, Davis, Sacramento, California, United States